CLINICAL TRIAL: NCT03188068
Title: Sirolimus Versus Sirolimus Plus Prednisolone for Kaposiform Hemangioendothelioma With Kasabach-Merritt Syndrome
Brief Title: Sirolimus Versus Sirolimus Plus Prednisolone for Kaposiform Hemangioendothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yi Ji, Principal Investigator, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-312; 81401606 (Other Grant/Funding Number: National Natural Science Foundation of China); 81400862 (Other Grant/Funding Number: National Natural Science Foundation of China); 2015SU04A15 (Other Grant/Funding Number: Excellent Youth Scholars of Sichuan University)
Record Dates: First submitted 2017-06-09; First posted 2017-06-15 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Kaposiform Hemangioendothelioma; Kasabach Merritt Phenomenon
Keywords: Kaposiform Hemangioendothelioma; Kasabach Merritt Phenomenon; Sirolimus; Prednisolone
MeSH Terms: conditions — Kaposiform Hemangioendothelioma; Kasabach-Merritt Syndrome | interventions — Sirolimus; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sirolimus (Active Comparator): Sirolimus was initiated at a dosage of 0.8 mg/m2 administered twice daily. Subsequently, the sirolimus dosage was adjusted monthly to achieve trough levels between 10 and 15 ng/mL.
  Interventions: Drug: Sirolimus
- Sirolimus plus prednisolone (Active Comparator): Sirolimus was initiated at a dosage of 0.8 mg/m2 administered twice daily. Subsequently, the sirolimus dosage was adjusted monthly to achieve trough levels between 10 and 15 ng/mL.
  Prednisolone was administered 2 mg/kg administered once daily. Should satisfactory clinical responses and hematologic stabilization ensue, prednisolone may be tapered and discontinued within the following 4-6 weeks.
  Interventions: Drug: Sirolimus; Drug: Prednisolone

INTERVENTIONS:
Drug: Sirolimus — Oral administration
  Other Names: Rapamycin
Drug: Prednisolone — Oral administered with sirolimus
  Arms: Sirolimus plus prednisolone

SUMMARY:
Kaposiform hemangioendothelioma (KHE) is a rare vascular neoplasm that occurs predominantly in infancy or early childhood. KHE has a nearly equal sex ratio. The annual incidence of KHE has been estimated at 0.071 per 100,000 children. KHE presents with intermediate-malignant and locally aggressive characteristics but without distant metastases.

This pilot trial studies sirolimus versus sirolimus plus pednisolone in treating patients diagnosed with kaposiform hemangioendothelioma (KHE) and Kasabach-Merritt phenomemon (KMP) that cannot be removed by surgery. The purpose of this study is to compare the efficacy and safety of orally administered sirolimus versus sirolimus plus pednisolone in the treatment of KHE associated with KMP.

DETAILED DESCRIPTION:
Kasabach-Merritt phenomemon (KMP) is a profound thrombocytopenia resulting from intralesional platelet trapping. It is now clear that KMP occurs with KHE and tufted angioma, not with infantile or congenital hemangiomas. KMP is typically associated with more aggressive lesions and poorer outcomes. Clinically significant KMP is a severe thrombocytopenia, generally below 30× 109/L. Severe thrombocytopenia may indicate a severer tumor, a progressive tumor, partially or totally insensitive to therapy. In addition to severe, persistent thrombocytopenia characteristic of KMP, patients often manifest elevated D-dimer and low fibrinogen. Coagulopathy in addition to thrombocytopenia is associated with more aggressive presentations and may indicate current infection or inflammation. Additionally, KMP may be complicated by severe anemia due to blood sequestration and intra-lesional hemorrhaging. KHE with KMP have notably high morbidity and mortality rates, resulting predominantly from rapid tumor growth and infiltration, compression or destruction of vital structures, and hemodynamic instability.

Consensus treatment guidelines from a multidisciplinary expert panel were published in 2013. Medical treatments with corticosteroids and/or vincristine have been recommended for the management of KHE. However, first-line treatment with corticosteroids is successful in only 10-27% of all cases, and treatment with vincristine is successful in 60-70% of patients. Moreover, vincristine monotherapy has not been confirmed to provide significant benefits in critically ill patients.

Sirolimus (also known as rapamycin) is an inhibitor of the mammalian target of rapamycin (mTOR). In recent studies, sirolimus was shown to be effective in patients with complex vascular anomalies, including KHE. Our multicenter, retrospective study demonstrated that oral sirolimus is an effective and safe option for the treatment of progressive KHE. Additionally, our data emphasized that the KHE treatment regimen should be tailored to individual patients and guided by specific clinical circumstances. In cases of severe Kasabach-Merritt phenomenon (KMP), sirolimus in combination with the short-term administration of prednisolone is recommended for controlling life-threatening conditions.

ELIGIBILITY:
Inclusion Criteria:

* Presenting a KHE with the following characteristics:

  1. Clinical features and histological findings consistent with progressive, non-resectable KHE associated with KMP.
  2. Patients must be 0 - 18 years of age at the time of study entry.
  3. Without functional impairment requiring treatment of corticosteroid.
* Organ function requirements:

  1 Adequate liver function:
  1. Total bilirubin less than or equal to 1.5 x upper limit of normal (ULN)for age, and
  2. ALT and AST less than or equal to 2.5 x upper limit normal (ULN) for age.

  2 Adequate renal function:
  1. 0-5 years of age maximum serum creatinine (mg/dL) of 0.8
  2. 6-10 years of age maximum serum creatinine (mg/dL) of 1.0
  3. 11-15 years of age maximum serum creatinine (mg/dL) of 1.2
  4. 16-18 years of age maximum serum creatinine (mg/dL) of 1.5
* Adequate bone marrow function: Absolute Neutrophil Count (ANC) greater than or equal to 1 x 10 to the ninth/Liter.
* Consent of parents (or the person having parental authority in families): Signed and dated written informed consent.

Exclusion Criteria:

* Allergy to sirolimus or other rapamycin analogues.
* Any known evidence of significant local or systemic uncontrolled infection, defined as receiving intravenous antibiotics at the time of randomization.
* Patients must not be known to be Human Immunodeficiency Virus positive or known immunodeficiency. Testing is not required unless a condition is suspected.
* Other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study (e.g. uncontrolled diabetes, uncontrolled hypertension, severe malnutrition, chronic liver or renal disease, active upper gastrointestinal tract ulceration).
* Impairment of gastrointestinal function or chronic gastrointestinal disease that may significantly alter the absorption of sirolimus.
* Patients who have a history of malignancy.
* Patients with an inability to participate or to follow the study treatment and assessment plan.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The changes of platelet counts | 2 months
  Platelet counts
The changes of fibrinogen levels | 2 months
  Fibrinogen levels
The changes in KHE volume | 6 and 12 months
  Response to therapy was measured by volumetric magnetic resonance imaging (MRI) analyses were performed at baseline and 6 and 12 months after treatment and were independently assessed by 2 radiologists. Changes in KHE size were classified as further growth (increase of ≥10%), no change (<10% increase and <10% decrease), partial involution (decrease of ≥10% and <75%), nearly complete involution (decrease of ≥75% and <100%), or complete involution (100%).
  Photographs of the mixed KHE were taken at months 0, 6 and 12 by a medical photographer.
The changes in the patient's symptoms and/or complications. | 6 and 12 months
  Improvement in the range of motion.

SECONDARY OUTCOMES:
Frequency of adverse events | 12 months
  Frequency of adverse events (e.g. gastrointestinal disorders, blood and lymphatic system disorders, metabolic disorders or other abnormal laboratory results, skin disorders and general disorders, etc.) collected by investigator and reported by parents. All adverse events were collected and graded according to Common Terminology Criteria for Adverse Events, version 4.0 (CTCAE v4.0). The causality of the adverse event was determined by the multidisciplinary staff and was classified as definitively not related, probably not related, possibly related, probably related, or definitively related. Any dose reductions, interruptions, or cessations enacted at the discretion of the investigators were recorded.
Change in blood biomarkers | 6 and 12 months
  Change in vascular endothelial growth factor (VEGF-A, C and D), IL-6, IL-8, angiopoietin 1 and 2. These parameters were measured via a series of correlative laboratory studies using blood samples.
Quality of life (QOL) in patients. | 12 months
  Pediatric Quality of Life Inventory (PedsQLTM) 4.0 Genetic Core Infant Scales (<2 years) or Pediatric Quality of Life Inventory (PedsQLTM) 4.0 Genetic Core Scales (2-18 years) were used.
Measuring the impact of KHE on family functioning. | 12 months
  PedsQLTM 4.0 Family Impact Module (FIM) was used.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ji, MD, PhD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ji Y, Chen S, Xiang B, Li K, Xu Z, Yao W, Lu G, Liu X, Xia C, Wang Q, Li Y, Wang C, Yang K, Yang G, Tang X, Xu T, Wu H. Sirolimus for the treatment of progressive kaposiform hemangioendothelioma: A multicenter retrospective study. Int J Cancer. 2017 Aug 15;141(4):848-855. doi: 10.1002/ijc.30775. Epub 2017 May 26. PMID 28486787
- [Background] Wang C, Li Y, Xiang B, Li F, Chen S, Li L, Ji Y. Successful Management of Pancreatic Kaposiform Hemangioendothelioma With Sirolimus: Case Report and Literature Review. Pancreas. 2017 May/Jun;46(5):e39-e41. doi: 10.1097/MPA.0000000000000801. No abstract available. PMID 28426496
- [Background] Reichel A, Hamm H, Wiegering V, Wiewrodt B, Neubauer H, Ernestus K, Winkler B. Kaposiform hemangioendothelioma with Kasabach-Merritt syndrome: successful treatment with sirolimus. J Dtsch Dermatol Ges. 2017 Mar;15(3):329-331. doi: 10.1111/ddg.12987. Epub 2017 Feb 21. No abstract available. PMID 28220608
- [Background] Alaqeel AM, Alfurayh NA, Alhedyani AA, Alajlan SM. Sirolimus for treatment of kaposiform hemangioendothelioma associated with Kasabach-Merritt phenomenon. JAAD Case Rep. 2016 Dec 5;2(6):457-461. doi: 10.1016/j.jdcr.2016.06.005. eCollection 2016 Nov. No abstract available. PMID 27981218
- [Background] Mahajan P, Margolin J, Iacobas I. Kasabach-Merritt Phenomenon: Classic Presentation and Management Options. Clin Med Insights Blood Disord. 2017 Mar 16;10:1179545X17699849. doi: 10.1177/1179545X17699849. eCollection 2017. PMID 28579853
- [Derived] Ji Y, Chen S, Zhou J, Yang K, Zhang X, Xiang B, Qiu T, Gong X, Zhang Z, Lan Y, Hu F, Kong F, Qiu Q, Zhang Y. Sirolimus plus prednisolone vs sirolimus monotherapy for kaposiform hemangioendothelioma: a randomized clinical trial. Blood. 2022 Mar 17;139(11):1619-1630. doi: 10.1182/blood.2021014027. PMID 35030255